CLINICAL TRIAL: NCT01106248
Title: An Open-Label, Multicenter, Single Arm QT Interval Prolongation Study of Eribulin Mesylate (E7389) in Patients With Advanced Solid Tumors
Brief Title: QT Interval Prolongation Study of Eribulin Mesylate (E7389) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-E044-110
Record Dates: First submitted 2010-04-14; First posted 2010-04-19 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-03

CONDITIONS: Advanced Solid Tumor
Keywords: tumor
MeSH Terms: conditions — Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eribulin Mesylate (Other)
  Interventions: Drug: Eribulin Mesylate

INTERVENTIONS:
Drug: Eribulin Mesylate — 1.4 mg/m^2 intravenous (IV) bolus given over 2-5 minutes on Days 1 and 8 every 21 days.

SUMMARY:
The purpose of this study is to assess whether eribulin mesylate (E7389) has an impact on the electrocardiogram (ECG) with focus on cardiac repolarization, as measured by QT/QTc interval as well as through a pharmacokinetic-pharmacodynamic (PK/PD) analysis.

DETAILED DESCRIPTION:
This is an open-label, multicenter, single arm QT Interval prolongation study of eribulin mesylate (E7389) in patients with advanced solid tumors.

ELIGIBILITY:
Personal history of unexplained syncope within the last year prior to entry

Inclusion Criteria:

1. Patients with histologically or cytologically confirmed advanced solid tumor that has progressed following standard therapy or for which no standard therapy exists (including surgery or radiation therapy).
2. Resolution of all chemotherapy or radiation-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy </= Grade 2 and alopecia.
3. Age >/= 18 years.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
5. Patients must have a sinus rhythm and QRS < 120msec.
6. Adequate renal function as evidenced by serum creatinine </= 2.0 mg/dL or calculated creatinine clearance >/= 40 mL/min per the Cockcroft and Gault formula.
7. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) >/= 1.5 x 10^9/L, hemoglobin >/= 10.0 g/dL (a hemoglobin <10.0 g/dL is acceptable if it is corrected by growth factor or transfusion), and platelet count >/= 100 x 10^9/L.
8. Adequate liver function as evidenced by bilirubin >/= 1.5 times the upper limits of normal (ULN) and alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) </= 3 x ULN (in the case of liver metastases </= 5 x ULN), unless there are bone metastases, in which case liver specific alkaline phosphatase must be separated from the total and used to assess the liver function instead of the total alkaline phosphatase.
9. Patients willing and able to comply with the study protocol for the duration of the study.
10. Written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria:

1. Patients who have received any of the following treatments within the specified period before start of treatment with eribulin mesylate:

   * Chemotherapy, radiation or biological therapy within three weeks
   * Hormonal therapy within one week
   * Any investigational drug within four weeks
2. Have had radiation therapy encompassing > 30% of bone marrow.
3. Have received prior treatment with mitomycin C or nitrosourea.
4. Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen.
5. Patients with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study. Any signs (e.g. radiologic) and/or symptoms of brain metastases must be stable for at least 4 weeks.
6. Patients with meningeal carcinomatosis.
7. Significant cardiovascular impairment (history of congestive heart failure > NYHA grade II, unstable angina or myocardial infarction within the past six months, or serious cardiac arrhythmia).
8. Patients with marked baseline prolongation of QT/QTc interval (QTc interval > 500 msec).
9. Patients with a history of additional risk factors for Torsades des pointes (e.g., heart failure, cardiac ischemia, recent Myocardial Infarction (MI), family history of Long QT Syndrome).
10. Patients with uncontrolled metabolic disorders (e.g hypokalemia, hypercalcemia and hypomagnesemia) at entry to the study.
11. Patients treated with antiarrythmic drugs or other medications that prolong the QT/QTc, that cannot be discontinued prior to entry into the study phase.
12. Patients with implantable pacemaker or automatic implantable cardioverter defibrillator (AICD).
13. .Bradycardia (defined as </= 50 beats/minute).
14. Personal history of unexplained syncope within the last year prior to entry into the study.
15. Patients with other significant disease or disorders that, in the Investigator's opinion, should exclude the patient from the study.
16. Patients who are receiving anti-coagulant therapy with warfarin or related compounds, other than for line patency, and cannot be changed to heparin-based therapy, are not eligible. If a patient is to continue on mini-dose warfarin, then the prothrombin time (PT) or international normalized ratio (INR) must be closely monitored.
17. Women who are pregnant or breast-feeding; women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test; women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator. Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
18. Severe/uncontrolled intercurrent illness/infection.
19. Patients with organ allografts requiring immunosuppression.
20. Patients with known positive HIV status.
21. Patients who have had a prior malignancy, other than carcinoma in situ of the cervix, or non-melanoma skin cancer, unless the prior malignancy was diagnosed and definitively treated >/= 5 years previously with no subsequent evidence of recurrence.
22. Patients with pre-existing neuropathy > Grade 2.
23. Patients with a hypersensitivity to halichondrin B and/or halichondrin B chemical derivative.
24. Patients who participated in a prior eribulin mesylate clinical trial.
25. Patients with pericardial effusion or pericardial metastases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jantien Wanders, MD, Study Director — Eisai Inc.
Locations (2):
- France (2):
  - Medicale, Dunkirk, *CS
  - Service d'Oncologie, Dunkirk, *CS

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 5 centers in France from Feb 2009 to Jul 2009.
Period: Overall Study
Arm/Group | Eribulin Mesylate
Started | 26
Completed | 23
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Administrative | 2

BASELINE CHARACTERISTICS:
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 55.9 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  France | 26

OUTCOME MEASURES:

1. Primary Outcome: Mean Time-matched, Baseline Corrected QTcF at Any Time Point Postdosing.
Description: The primary endpoint is mean time-matched, baseline corrected QTcF at any time point postdosing. This was to determine the effect of eribulin on cardiac repolarization as measured by QT/QTc interval.
Time Frame: 48 hours postdose after Day 1 and after Day 8
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 26
msec
  Postdosing Day 1 | 2 (12.3)
  Postdosing Day 8 | 11 (18.7)

2. Secondary Outcome: Pharmacokinetic Profile of Eribulin Mesylate: Observed Maximal Plasma Concentration (Cmax)
Description: Pharmacokinetic profile of eribulin mesylate (Cmax).
Time Frame: Days 1 and 8
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 26
ng/mL
  Day 1 | 516.5 (137.91)
  Day 8 | 502.4 (138.31)

3. Secondary Outcome: To Assess Best Overall Response Using RECIST Criteria in Patients With Measurable Disease.
Time Frame: 21 day cycle
Reporting Status: Not Posted

4. Secondary Outcome: To Further Explore the Safety and Tolerability of Eribulin Mesylate When Administered on Days 1 and 8 of a 21-day Cycle in Patients With Solid Tumors.
Time Frame: 21 day cycle
Reporting Status: Not Posted

5. Secondary Outcome: Pharmacokinetic Profile of Eribulin Mesylate: Time to Maximum Observed Plasma Concentration (Tmax).
Description: Pharmacokinetic profile of eribulin mesylate (tmax).
Time Frame: Days 1 and 8
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: hours
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 26
hours
  Day 1 | 0.08 [0.07 to 0.25]
  Day 8 | 0.08 [0.05 to 0.25]

ADVERSE EVENTS:
Arm/Group | Eribulin Mesylate
Serious Adverse Events (participants affected / at risk) | 11/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=26)
General Physical Health Deterioration (General disorders) | 5
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 2
Non-Cardiac Chest Pain (General disorders) | 1
Vomting (Gastrointestinal disorders) | 2
Subileus (Gastrointestinal disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 3
Bacteremia (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Diplopia (Eye disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Weight Decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=26)
Constipation (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 9
Abdominal Pain (Gastrointestinal disorders) | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Bezoar (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Fecal Incontinence (Gastrointestinal disorders) | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Esophageal Pain (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 14
Pyrexia (General disorders) | 9
Fatigue (General disorders) | 5
General Physical Health Deterioration (General disorders) | 5
Peripheral Edema (General disorders) | 4
Mucosal Inflammation (General disorders) | 2
Chills (General disorders) | 1
Malaise (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 16
Anemia (Blood and lymphatic system disorders) | 12
Leukopenia (Blood and lymphatic system disorders) | 10
Lymphopenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Paratracheal Lymphadenopathy (Blood and lymphatic system disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 3
Parasthesia (Nervous system disorders) | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Intracranial Pressure Increased (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraparesis (Nervous system disorders) | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 1
Tongue Paralysis (Nervous system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 11
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Oral Herpes (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Bacteremia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Catheter Related Infection (Infections and infestations) | 1
Fungal Skin Infection (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Alanine Aminotransferase Increased (Investigations) | 3
Aspartate Aminotransferase Increased (Investigations) | 3
Weight Decreased (Investigations) | 3
Gamma Glutamyltransferase Increased (Investigations) | 2
Alanine Aminotransferase Decreased (Investigations) | 1
Blood Alkaline Phosphatase Increased (Investigations) | 1
Blood Bilirubin Increased (Investigations) | 1
Gamma Glutamyltransferase Decreased (Investigations) | 1
Weight Increased (Investigations) | 1
Insomnia (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 2
Confusional State (Psychiatric disorders) | 2
Agitation (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Urinary Retention (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Tinnitis (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hepatic Pain (Hepatobiliary disorders) | 2
Cholestasis (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Conjunctivitis (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Hypotension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No